CLINICAL TRIAL: NCT03368495
Title: Immunogenicity of Co-administered Yellow Fever and Measles, Mumps, and Rubella (MMR) Vaccines in Children Under 2 Years Old in Argentina
Brief Title: Immunogenicity of Co-administered Yellow Fever and Measles, Mumps, and Rubella (MMR) Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alba Maria Ropero (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Public Health, Argentina (Other Government)
Responsible Party: Sponsor-Investigator, Alba Maria Ropero, Regional Advisor, Immunization Unit, Pan American Health Organization
Organization: Pan American Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAHO-2014-07-0011
Record Dates: First submitted 2017-11-21; First posted 2017-12-11 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Vaccine Response Impaired
Keywords: yellow fever vaccine; MMR vaccine; immunogenicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-administration of MMR/YF (Experimental): Participants randomized to this arm will receive both MMR and yellow fever vaccines on Day 0.
  Interventions: Biological: Co-administration of MMR/YF
- MMR followed by YF (Active Comparator): Participants randomized to this arm will receive MMR vaccine on Day 0 followed by yellow fever vaccine on Day 28.
  Interventions: Biological: MMR followed by YF
- YF followed by MMR (Active Comparator): Participants randomized to this arm will receive YF vaccine on Day 0 followed by MMR vaccine on Day 28.
  Interventions: Biological: YF followed by MMR

INTERVENTIONS:
Biological: Co-administration of MMR/YF — Both MMR & yellow fever vaccines administered on Day 0.
  Arms: Co-administration of MMR/YF
Biological: MMR followed by YF — MMR vaccine administered on Day 0 and yellow fever vaccine administered on Day 28.
  Arms: MMR followed by YF
Biological: YF followed by MMR — Yellow fever vaccine administered on Day 0 and MMR vaccine administered on Day 28.
  Arms: YF followed by MMR

SUMMARY:
This study evaluates seroconversion against measles, mumps, rubella and yellow fever following vaccination. One-third of children will receive both yellow fever and measles, mumps, and rubella (MMR) vaccines on the same day; one- third of children will receive MMR vaccine at enrollment followed by yellow fever vaccine 4 weeks later; one-third of children will receive yellow fever vaccine at enrollment followed by MMR vaccine 4 weeks later.

DETAILED DESCRIPTION:
The World Health Organization (WHO) and the Pan American Health Organization recommend that yellow fever and measles, mumps and rubella (MMR) vaccines be administered on the same day or at least 4 weeks apart to prevent interference between live vaccines. In 2011 a Brazilian study demonstrated lower seroconversion against yellow fever, rubella, and mumps when the two vaccines were administered on the same day compared with administering them separately. WHO urged that additional studies be conducted to examine this issue.

This Phase IV study aims to determine if seroconversion against measles, mumps, rubella, and yellow fever after administration of MMR and yellow fever vaccines on the same day is non-inferior to seroconversion after sequential administration 28 days apart in health 12-month old children.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 24 months at the time of enrollment
* Healthy child, determined by clinical history
* Availability to do study visits and blood sampling on days 28 + 7 and 56 + 14
* Informed consent signed by parents

Exclusion Criteria:

* Previous vaccination against yellow fever, measles, mumps, or rubella
* History of yellow fever, measles, mumps or rubella
* Contraindication for any of the study vaccines: yellow fever vaccine or triple viral vaccine, including:

  1. Allergy to eggs, gelatin, or neomycin
  2. Weakened immunological function, including HIV infection, primary immunodeficiencies, having received immunosuppressive doses of oral or injectable corticosteroids (or equivalent), having received immunomodulators or chemotherapeutic agents
  3. Thymus disease
  4. Serious illness/fever (mild illness without fever is not an exclusion criterion)
* Administration of immunoglobulins or other blood derivative within 6 months of enrollment in the study or during the study

  a. Exception: children with a history of Kawasaki disease who received gammaglobulin cannot be enrolled if they received it in the previous 11 months.
* Administration of any other attenuated viral vaccine (i.e., for chickenpox) in the month prior to enrollment, or if the administration of any other attenuated viral vaccine is expected during the study (up to 3 months)
* Not being available for the entire study period (up to 3 months), or not able to make the scheduled visits or complete the study procedures
* Participating in another clinical drug trial of a drug, vaccine, or medical device
* Any condition that, in opinion of the study staff, represents a health risk to the participant or interferes with the evaluation of the response to the vaccine (i.e., children in percentile ≤ 3 in the height/weight tables will be considered undernourished and cannot be selected)

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 851 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Seroconversion after yellow fever vaccination using the plaque reduction neutralization test (PRNT). | 28-35 days post-vaccination
  PRNTs will be used to measure antibody titers for yellow fever.
Seroconversion after MMR vaccination using the ELISA method. | 28-35 days post-vaccination.
  The ELISA method will be used to measure antibody titers for measles, mumps, and rubella.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Biscayart, MD, Principal Investigator — Minsterio de Salud de la Nacion, Argentina
Locations (4):
- Argentina (4):
  - SAMIC Eldorado Hospital, Eldorado, Misiones Province
  - SAMIC Obera Hospital, Oberá, Misiones Province
  - Favoloro Hospital, Posadas, Misiones Province
  - IPS Hospital, Posadas, Misiones Province

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vizzotti C, Harris JB, Aquino A, Rancano C, Biscayart C, Bonaventura R, Pontoriero A, Baumeister E, Freire MC, Magarinos M, Duarte B, Grant G, Reef S, Laven J, Wannemuehler KA, Alvarez AMR, Staples JE. Immune response to co-administration of measles, mumps, and rubella (MMR), and yellow fever vaccines: a randomized non-inferiority trial among one-year-old children in Argentina. BMC Infect Dis. 2023 Mar 17;23(1):165. doi: 10.1186/s12879-023-08114-1. PMID 36932346